CLINICAL TRIAL: NCT01440491
Title: Effect of Orientation Through a Booklet of Exercise in Patients With Low Back Pain
Brief Title: Orientation Booklet for Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rioko Kimiko Sakata, Pain Clinic Director, Federal University of São Paulo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP1871/07
Record Dates: First submitted 2011-09-13; First posted 2011-09-26 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2008-01

CONDITIONS: Low Back Pain
Keywords: low back pain; exercise; booklet
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- physiotherapy orientated (Other): G1 patients were orientated by the physiotherapist during the performance of physiotherapy exercises, using the booklet
  G2 received the booklet to self perform the physiotherapy exercises
  Interventions: Other: Physiotherapy exercise

INTERVENTIONS:
Other: Physiotherapy exercise — once a day, during 15 minutes, for 12 weeks
  Other Names: Exercise therapy

SUMMARY:
The aim of this study was to evaluate the effect of exercises performed under monitoring of the physiotherapist and self performed at home by reading the booklet of exercise orientation for patients with nonspecific low back pain.

A prospective and randomized trial was performed in 44 patients. G1 patients received a physiotherapist orientation, and G2 patients received the booklet of exercise to self perform the exercises. Pain intensity by Visual Analogue Scale (VAS), and quality of life by SF-36 were measured before.

Results: Pain intensity was lower in G1 than in G2 after 6 and 12 weeks. Quality of life was better in G1.

The exercises under orientations of the physiotherapist promoted best effect than self performed exercises .

DETAILED DESCRIPTION:
After approval by the Ethics Committee and signing a consent form, a prospective, randomized trial was performed in 44 patients with chronic nonspecific low back pain (lasting longer than 3 months), pain intensity greater than 3 by visual analogue scale and age > 18 years. Patients with renal and gastrointestinal disease, simultaneously submitted to another type of physical therapy, cognitive impairment, and pregnant women were excluded.

All patients received an exercise booklet which consisted of stretching and strengthening of muscles. G1 patients were orientated by the physiotherapist during the performance of exercises once a week, using the booklet, and the patients in G2 (n=22) received the booklet to self perform the exercises without orientation of the physiotherapist. Everyone should perform the exercises once a day at home.

Pain intensity by VAS, and quality of life by SF-36 were measured before the start of treatment (T0), after 6 (T6) and 12 (T12) weeks. Side effects were recorded. Acetaminophen (up to 4 g / day) could be used as necessary.

The sample size was provided by SAS 8.0, SPSS 15.0 program. To detect difference in pain intensity of 3 between the groups by VAS, with 95% of power (estimated SD= 2.0), when the alpha level is set at 0.05, the sample should be of 16. The program used for statistical analysis was SAS 8.0, SPSS 15.0. The tests used were Student's T to compare age of patients, chi-square to compare gender and analgesic complementation, and Mann Whitney test for pain intensity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* chronic nonspecific low back pain (lasting longer than 3 months),
* pain intensity greater than 3 by visual analogue scale and age > 18 years

Exclusion Criteria:

* Patients with renal and gastrointestinal disease,
* simultaneously submitted to another type of physical therapy,
* cognitive impairment, and
* pregnant women were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Pain | 12 weeks
  Pain intensity was measured by VAS, and quality of life by SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, MD, PhD, Study Director — Universidade Federal de São Paulo